CLINICAL TRIAL: NCT02440425
Title: Phase 2 Trial of Dose Dense (Weekly) Paclitaxel With Pembrolizumab (MK-3475) in Platinum Resistant Recurrent Ovarian Cancer
Brief Title: Dose Dense Paclitaxel With Pembrolizumab (MK-3475) in Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18207
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer
Keywords: platinum resistant; recurrent; persistent; epithelial; ovarian; fallopian tube; primary peritoneal; carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence; Carcinoma | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy (Experimental): Combination Therapy: Pembrolizumab (experimental use) and Paclitaxel (standard use). All trial treatments will be administered on an outpatient basis. One cycle equals 21 days. The first cycle is 28 days with Pembrolizumab given on day 8 in order to determine paclitaxel tolerance.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab: 200 mg, every (Q) 3 weeks, via intravenous (IV) infusion, until progression or toxicity (or up to 24 months). The first cycle will begin on day 8.
  Other Names: MK-3475; KEYTRUDA®
Drug: Paclitaxel — Paclitaxel: 80 mg/m^2, Q week for 3 weeks, via IV infusion, until progression or toxicity (or complete response if at least 6 cycles, at the discretion of the investigator and participant). Cycle 1 will have an extra lead in week (4 weeks total) with Paclitaxel only on week 1.
  Other Names: Taxol; Onxal

SUMMARY:
The purpose of this study is to find out if the combination of Paclitaxel once per week with Pembrolizumab once every 3 weeks will help participants with this disease. Researchers want to find out the effectiveness of the drug combination to improve the delay of cancer progression or death and compare it to historical data for weekly paclitaxel alone, and assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmation of the histologic diagnosis of high-grade (grade 2-3) epithelial, non-mucinous, non-borderline, ovarian, fallopian tube, or primary peritoneal carcinoma. May be based on original pathology report or review of original slides.
* Willing and able to provide written informed consent/assent and authorization
* ≥ 18 years of age on day of signing informed consent
* Disease must have been persistent or have recurred within 6 months of prior platinum therapy. Disease may not have progressed during prior platinum therapy (i.e., refractory).
* Have measurable disease or detectable (non-measureable) disease
* Measurable disease: must have at least one "target lesion" to be used to assess response on this protocol.
* Prior Therapy:

  * Have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents (biologic/ targeted) or extended therapy administered after surgical or non-surgical assessment. If patients were treated initially with paclitaxel for their primary disease, this can have been given weekly or every 3 weeks. The most recent therapy and any therapies subsequent to initial therapy, however, cannot have contained weekly paclitaxel. If the immediate prior (most recent therapy) is the initial therapy, it may not have been with weekly paclitaxel.
  * Allowed to receive (not required to receive), 2 additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum regimen. Treatment with weekly paclitaxel for recurrent or persistent disease is NOT allowed.
  * Allowed to receive(not required to receive), non-cytotoxic (biologic/targeted) therapy as part of their primary treatment regimen. Allowed to receive (not required to receive), non-cytotoxic (biologic/targeted) therapy as part of their treatment for recurrent or persistent disease and/or as treatment for recurrent or persistent disease. If non-cytotoxic (biologic/targeted) therapy is given alone (i.e., not in combination with cytotoxic chemotherapy) it will NOT count as a prior regimen.
* Have tissue from an archival tissue sample that has been identified and confirmed as available for study, or newly obtained core or excisional biopsy of a tumor lesion
* Have received 1 prior regimen must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2. If have received 2 or 3 prior regimens, must have an ECOG Performance Status of 0 or 1.
* Adequate organ function as defined in the protocol
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy: Should be free of active infection requiring antibiotics (with exception of uncomplicated UTI); Any hormonal therapy directed at the malignant tumor must be discontinued at least 2 weeks prior to registration (continuation of hormone replacement therapy is permitted); Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted and immunologic agents, must be discontinued at least 2 weeks prior to registration and at least 3 weeks before day 1 on trial.
* Women of Childbearing Potential (WOCBP): Negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* WOCBP willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.

Exclusion Criteria:

* Have low-grade or non-epithelial cancers, mucinous cancers, and/or borderline low-malignant potential cancers
* Currently participating in/have participated in a study of an investigational agent or is or has been using an investigational device within 4 weeks of the first dose of treatment
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to prior therapies
* Had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: If received major surgery, must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* History of other invasive malignancies (with exception of non-melanoma skin cancer and or in situ cancers that have undergone potentially curative therapy) are excluded if there is any evidence of other malignancy being present within the last 3 years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last 3 years are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last 3 year. May have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease.
* History of synchronous endometrial cancer unless all of the following conditions are met: Stage not greater than I-A (FIGO 2010 staging criteria); no more than superficial myometrial invasion (<50%), without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO Grade 3 lesions and it has been greater than 3 years since diagnosis and there have been no recurrences.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment..
* Evidence of interstitial lung disease, any active, non-infectious pneumonitis, or known active tuberculosis
* An active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating physician or the principal or study investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Known active Hepatitis B or Hepatitis C
* Received a live vaccine within 30 days prior to the first dose of trial treatment
* Peripheral neuropathy Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher
* Known hypersensitivity to pembrolizumab or any of its excipients
* Known hypersensitivity to paclitaxel
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wenham, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Duke University, Durham, North Carolina
  - VCU Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 42
Completed | 37
Not Completed | 5
Not completed — Death likely due to disease progression | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Adverse Event/Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Number of participants who received at least one dose of study drugs.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 6 Months
Description: 6-month progression-free survival of the combination of weekly paclitaxel with pembrolizumab (MK-3475) for those patients who received treatment and were evaluable (had one response assessment scan by RECIST 1.1) . 6-month PFS: The proportion of patients at 6 months alive without progressive disease. Progressive Disease (PD): Sum of the longest diameters (SLD) increased by at least 20% from the smallest value on study (including baseline, if that is the smallest).
Time Frame: 6 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 37
percentage of participants | 58.6 [41.0 to 72.7]

2. Primary Outcome: Occurrence of Adverse Events
Description: Safety of the combination of paclitaxel weekly with pembrolizumab every 3 weeks (Q3W). Serious Adverse Events and Adverse Events will be reported in that Results Data section, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.0.
Time Frame: 2 years, 6 months
Population: All participants who received at least one dose of study drugs.
Measure: Number; unit: Events
Arm/Group | Combination Therapy
Number analyzed (Participants) | 42
Events
  SAEs related to study treatment | 28
  AEs related to study treatment | 573

3. Secondary Outcome: Response Rate (RR)
Description: Proportion of participants who respond to the regimen by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. RECIST v1.1: Complete Response (CR) - Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis. Partial Response (PR) - At least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. RR=CR + PR.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 37
percentage of participants | 51.4 [34.4 to 68.1]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR: The percentage of participants complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents. Stable Disease (SD) - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. DCR=CR + PR + (SD x 2 mo.)
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 37
percentage of participants | 86.5 [75.5 to 97.5]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response in months. DOR= Duration from first observation of partial response to the time of disease progression.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 37
months | 8.8 [4.4 to 13.0]

6. Secondary Outcome: Median Overall Survival (OS)
Description: OS: The time from randomization until death from any cause.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 37
months | 26.3 [13.4 to 35.1]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from Day 1 of treatment through Day 90 after treatment, 4 years, 6 months. All participants who received at least one dose of study drug are included.
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 25/42
Serious Adverse Events (participants affected / at risk) | 21/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=42)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Edema (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cough (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Related to diabetes and dehydration
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (5)
Fever (General disorders) | 3 (6)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1) — gram positive alpha hemolytic strep
Chills (General disorders) | 1 (1)
Infections and Infestations-Other (Infections and infestations) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=42)
Fatigue (General disorders) | 31 (51)
Edema limbs (General disorders) | 23 (34)
Fever (General disorders) | 11 (17)
Pain (General disorders) | 11 (12)
Non-cardiac chest pain (General disorders) | 8 (9)
Flu-like symptoms (General disorders) | 7 (7)
Chills (General disorders) | 6 (6)
Infusion related reaction (General disorders) | 4 (4)
Edema face (General disorders) | 3 (3)
Malaise (General disorders) | 2 (2)
Edema trunk (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 38 (205)
Leukocytosis (Blood and lymphatic system disorders) | 9 (23)
Investigations - Other (Investigations) | 29 (103)
Neutrophil count decreased (Investigations) | 27 (100)
White blood cell count decreased (Investigations) | 23 (121)
Lymphocyte count decreased (Investigations) | 22 (104)
Alkaline phosphatase increased (Investigations) | 16 (34)
Aspartate aminotransferase increased (Investigations) | 14 (18)
Activated partial thromboplastin time prolonged (Investigations) | 13 (26)
Alanine aminotransferase increased (Investigations) | 12 (14)
Platelet count decreased (Investigations) | 11 (17)
Creatinine increased (Investigations) | 4 (10)
INR increased (Investigations) | 4 (4)
CPK increased (Investigations) | 2 (4)
Weight gain (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 18 (43)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (35)
Anorexia (Metabolism and nutrition disorders) | 14 (16)
Hyponatremia (Metabolism and nutrition disorders) | 12 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (14)
Hypokalemia (Metabolism and nutrition disorders) | 10 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (38)
Diarrhea (Gastrointestinal disorders) | 19 (35)
Vomiting (Gastrointestinal disorders) | 18 (27)
Bloating (Gastrointestinal disorders) | 13 (19)
Constipation (Gastrointestinal disorders) | 13 (14)
Abdominal pain (Gastrointestinal disorders) | 11 (15)
Abdominal distension (Gastrointestinal disorders) | 5 (7)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 (5)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Ascites (Gastrointestinal disorders) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8 (14)
Nail loss (Skin and subcutaneous tissue disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Bulbous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (21)
Peripheral motor neuropathy (Nervous system disorders) | 9 (12)
Dizziness (Nervous system disorders) | 8 (10)
Dysgeusia (Nervous system disorders) | 3 (3)
Parasthesia (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness, lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 8 (10)
Nail infection (Infections and infestations) | 4 (4)
Infections and infestations - Other (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 9 (41)
Hypotension (Vascular disorders) | 6 (8)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (9)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 4 (6)
Proteniuria (Renal and urinary disorders) | 4 (8)
Renal and urinary disorders -Other (Renal and urinary disorders) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 6 (6)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (7)
Hyperthyroidism (Endocrine disorders) | 3 (4)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Endocrine disorders - Other (Endocrine disorders) | 1 (2)
Eye disorders - Other (Eye disorders) | 3 (4)
Watering eyes (Eye disorders) | 2 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hepatobiliary disorders -Other (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Primary outcome only incorporated patients who received treatment & completed first RECIST 1.1 response assessment. Does not reflect an intent-to-treat population.

All patients enrolled & received one dose of drug were included for safety analysis.

Although patients had a recurrence of cancer within 6 months of a platinum drug ("platinum-resistant"), 43% of patients were enrolled on study >6 months from last platinum-based therapy (including maintenance) & 16.2% were greater than 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study may be presented at scientific meetings by any of the study investigators with the approval of the Sponsor and also allowing time for prior review by Merck. Intent to submit should be made no later than 4 weeks before a submission is due, and a copy of an abstract or presentation should be submitted no later than 3 weeks prior to finalization or submission to allow time to review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT02440425/Prot_SAP_000.pdf